CLINICAL TRIAL: NCT03534427
Title: The Effects of a 12-Week Jump Rope Exercise Training Program on Arterial Stiffness, Vasodilating and Vasoconstricting Factors, Inflammatory Markers, and Body Composition in Prehypertensive Adolescent Girls
Brief Title: The Effects of a Jump Rope Exercise Program on Vascular Health, Inflammatory Markers in Prehypertensive Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PusanNU1
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Results first posted 2019-08-14 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Prehypertension; Blood Pressure; Abdominal Obesity; Adiposity
Keywords: arterial stiffness; endothelin-1; c-reactive protein; adiposity; exercise; jump rope
MeSH Terms: conditions — Prehypertension; Obesity, Abdominal; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: exercise intervention group, control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No exercise intervention
- Jump rope exercise intervention (Experimental): The jump rope exercise program was performed for 50 minutes with 5 minutes of warm-up and cool-down per day, 5 times a week for 12 weeks. The program consisted of various main jump rope exercises (1 line 2 jump, jumping feet together, running jumping, open side jump, open back and forth jump, rock paper scissor jump). The warm-up and cool down consisted of static stretching, walking, and jogging. Intensity of exercise was gradually increased from 40-50% heart rate reserve (HRR) in weeks 1-4 and to 60-70% HRR in weeks 9-12. Each training session was supervised by the researchers. Every subject wore a heart rate monitor during the whole training session in order to maintain the designated training intensity.
  Interventions: Other: Jump rope exercise intervention

INTERVENTIONS:
Other: Jump rope exercise intervention — 12-week jump rope exercise program
  Arms: Jump rope exercise intervention

SUMMARY:
The purpose of this study was to examine the impact of a 12-week jump rope exercise program on blood pressure, arterial stiffness, vasodilating and vasoconstricting factors, inflammatory markers, and body composition in prehypertensive adolescent girls. Forty prehypertensive adolescent girls participated in this study. The girls were randomly divided into the jump rope exercise intervention group (EX, n=20) and control group (CON, n=20). The EX group performed a jump rope training program at 40-70% of their heart rate reserve (HRR) 5 days/week for 12 weeks (sessions 50 minutes in duration). The CON group did not participate in any structured or unstructured exercise protocol. Blood pressure, arterial stiffness, plasma nitrate/nitrite levels, endothelin-1, C-reactive protein, and body composition were measured before and after the 12-weeks study.

ELIGIBILITY:
Inclusion Criteria:

* prehypertensive
* sedentary (no regular exercise training or physical activity within the last year)
* no weight loss diet during the last six months

Exclusion Criteria:

* pregnancy
* chronic disease
* daily medication use (including antioxidants and weight loss supplements)

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2011-06-05 (Actual); Primary Completion 2012-02-10 (Actual); Study Completion 2012-03-21 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Jump Rope Exercise Intervention
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Jump Rope Exercise Intervention | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.2) | 15.3 (0.9) | 15.1 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 20 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 20 | 20 | 40
Arterial stiffness [Mean (Standard Deviation); unit: m/s] | 8.2 (0.5) | 8.2 (1) | 8.2 (0.8)
Endothelin-1 [Mean (Standard Deviation); unit: umol/mL] | 0.41 (0.21) | 0.37 (0.21) | 0.40 (0.21)
Body mass [Mean (Standard Deviation); unit: kg] | 68 (8) | 69 (9.4) | 68.5 (8.7)
Height [Mean (Standard Deviation); unit: cm] | 161 (3) | 160 (3) | 160.5 (3)
Waist circumference [Mean (Standard Deviation); unit: cm] | 85.3 (4) | 86.4 (4) | 85.9 (4)
Body Fat [Mean (Standard Deviation); unit: percent] | 32.7 (3.2) | 33.8 (3.6) | 33.3 (3.4)
Lean Body Mass [Mean (Standard Deviation); unit: kg] | 43.7 (4.2) | 44.9 (4.5) | 44.3 (4.3)
Nitrate/Nitrite Levels [Mean (Standard Deviation); unit: umol] | 53.3 (4.3) | 54.5 (5.1) | 53.9 (4.7)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] | 0.5 (0.3) | 0.5 (0.4) | 0.5 (0.4)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 126 (4.2) | 126 (3.3) | 126 (3.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 82 (2) | 82 (0.4) | 82 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Arterial Stiffness
Description: Arterial stiffness was measured as measurement of brachial to ankle pulse-wave velocity. This indicates peripheral arterial stiffness, as it measures how quickly a pulse wave propagates from one point to another.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
m/s | 8.1 (0.2) | 7.4 (0.2)

2. Primary Outcome: Endothelin-1
Description: Levels of Endothelin-1 in blood were measured by Endothelin-1 enzyme immunoassay kit.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: umol/mL
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
umol/mL | 0.4 (0.31) | 0.38 (0.33)

3. Primary Outcome: Body Mass
Description: Body mass was measured to nearest 0.1 kg.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
kilograms (kg) | 70 (8.9) | 66 (7.3)

4. Primary Outcome: Height
Description: Height was measured to nearest 1 cm.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
cm | 162 (4) | 161 (3)

5. Primary Outcome: Waist Circumference
Description: Waist circumference was measured at midpoint between the lower rib and the iliac crest at the end of a normal expiration using a tape measure.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
cm | 84.4 (5.2) | 80.1 (4.8)

6. Primary Outcome: Body Fat
Description: Percent body fat (%) was determined using a bioelectrical impedance-meter.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
percent | 33.5 (3.7) | 30.2 (3.1)

7. Primary Outcome: Lean Body Mass
Description: Lean body mass (kg) was determined using a bioelectrical impedance-meter.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
kilograms (kg) | 42.8 (6.5) | 45.9 (6.7)

8. Primary Outcome: Nitrate/Nitrite Levels
Description: Nitrate and nitrite levels were assayed using a Griess assay kit.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: umol
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
umol | 53.5 (5.2) | 57.2 (5.2)

9. Primary Outcome: C-reactive Protein
Description: C-reactive protein was assessed using an enzyme immunoassay assay kit
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
mg/L | 0.7 (0.4) | 0.2 (0.1)

10. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured in duplicate using an automated sphygmomanometer. The average of the two was recorded as the resting blood pressure.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
mmHg | 127 (5.3) | 120 (2.1)

11. Primary Outcome: Diastolic Blood Pressure
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Jump Rope Exercise Intervention
Number analyzed (Participants) | 20 | 20
mmHg | 84 (1.9) | 80 (2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Group | Jump Rope Exercise Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03534427/Prot_SAP_000.pdf